CLINICAL TRIAL: NCT02865889
Title: Cost-Effectiveness and Patients Satisfaction of Conventional vs Robotic-Assisted Laparoscopy in Gynecologic Oncologic Indications
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: STIC COELCO
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: UTERINE CERVICAL NEOPLASMS; ENDOMETRIAL NEOPLASMS
Keywords: laparoscopic surgery; Uterine Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Uterine Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Uterine oncologic Indications for surgery
  Interventions: Procedure: Laparoscopy in Gynecologic Oncologic Indications; Procedure: Conventional surgery (abdominal radical surgery)

INTERVENTIONS:
Procedure: Laparoscopy in Gynecologic Oncologic Indications
Procedure: Conventional surgery (abdominal radical surgery)

SUMMARY:
Laparoscopic surgery is gaining currency in the field of oncologic care, particularly for colorectal and gynecologic cancers. This innovation could be used either for staging purpose and therefore could steer global therapeutic options or for surgical management only.

Increase knowledge and skills lead to an increase in the number and rate of the women this innovation could be offered. The project team observed a shift from traditional surgical management (abdominal radical surgery) towards laparoscopic with a focus on lymphadenectomy.

This innovation however increases some costs (the surgical stage) but decrease some others (the post surgical stage).

Foreseeing the pace of the dissemination needs to have objective and reliable data about who had access to laparoscopic surgery and who didn't (and why) and accurate assessment of related costs.

This program will focus on uterine cancer (both cervix and corpus).

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Endometrial or cervical cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endometrial and cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2008-09; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cost comparison between Conventional vs Robotic-Assisted Laparoscopy | 2 years
  The following costs were included:Equipment costs,Instrument costs,Operating room costs,Hospital stay
Comparison of the effectiveness of procedures (Conventional vs Robotic-Assisted Laparoscopy) | 2 years
  Comparison of the effectiveness of procedures will take into account conversion rate, complications rate, metastatic and pelvic relapse

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lambaudie, MD,PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du Rhône, France